CLINICAL TRIAL: NCT02055235
Title: Pain Processing and Pain Control in Experienced Yoga Practitioners
Brief Title: Study of Pain Processing in Experienced Yoga Practitioners
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140054; 14-AT-0054
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2016-10-12

CONDITIONS: Pain
Keywords: Brain; Pain; Yoga
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Different people perceive the same pain differently. Mood, attention, stress, and personality affect how we feel pain. Researchers want to know whether people who do yoga perceive pain differently than people who do not practice yoga, meditation, or martial arts. They also want to study if cortisol, a stress hormone, relates to pain or brain differences.

Objective:

- To study the effects of yoga on the body s stress response, pain perception, and the brain s structure and pain response.

Eligibility:

* Right-handed adults 30 years and older who practice yoga regularly.
* Healthy right-handed volunteers 30 years and older who do at least mild exercise but no yoga or martial arts.

Design:

* Visit 1: Participants will be screened with medical history and physical exam. They will have blood and urine tests and electrocardiogram to measure heart activity.
* At home, participants will wear a heart monitor for 1 day and collect 5 saliva samples daily for seven days.
* Visit 2: Participants will undergo tests in a chair or in a mock MRI machine. They will lie on a table that slides into a cylinder.
* A heating device will be placed on their leg and heated periodically for few seconds at a time.
* They will give saliva samples.
* Heart rate, respiration, etc. will be monitored.
* They will fill out questionnaires.
* Visit 3: Participants will answer questions and repeat Visit 2 tests. Tests will be done in the real MRI machine. The scanner makes loud knocking sounds. Participants will get earplugs. Participants will be in the scanner about 1 hour with a coil over their head.

DETAILED DESCRIPTION:
Objective: Pain perception is characterized by substantial differences between individuals. We recently showed that a group of experienced yogis tolerated pain much longer than matched controls. To tolerate pain yogis reported using strategies involving interoceptive awareness and parasympathetic activation while nearly all controls did not. Yogis had more gray matter in multiple brain regions, but only mid-insular gray matter correlated with pain tolerance. They also had higher left intra-insular white matter connectivity than controls. Given that autonomic integration occurs in the mid-insula, these observed insular adaptations could be related to successful pain affect regulation mediated by increased interoceptive processing and parasympathetic regulation. Our findings are consistent with a recent theory suggesting that yoga s benefits are achieved by reducing allostatic load in stress response systems ( wear and tear on the body ), thus restoring optimal homeostasis. Specifically, the beneficial effects of yoga on many conditions, including chronic pain, may be attributable to increased parasympathetic activation. Indeed, all the conditions benefiting from yoga practice are exacerbated by stress and exhibit a high sympathetic/parasympathetic balance, as measured by low heart rate variability (HRV). Increased sympathetic activity is known to increase hypothalamo-pituitary-adrenal (HPA) axis function. Additionally, it has been proposed that people respond to uncertainty by activating the sympathetic nervous system, and that this default response is related to the well-known negativity bias, the tendency to prioritize negative information over positive. Yoga teaches a more neutral appraisal of the world which might be a better adaptive response to uncertainty not involving as much sympathetic activation and requiring less energy from the organism than prioritizing negative information in a reactive way. This should promote a better control over stressful events including pain. Thus, the proposed studies will first pilot the psychophysical procedures before proceeding to the full study testing general hypothesis that the differences in pain processing and the related neurostructural and neurophysiological differences expected to be found in experienced yogis are related to more flexible autonomic and HPA axis control. We will also document personality traits, including pain-related behaviors, and mental states associated with the observed differences.

Study population: In the pilot sub-study 19 experienced yogis will be compared to 19 healthy volunteers who will serve as controls. The full protocol will include 49 participants per group.

Design: A pilot sub-study will be followed by the full cross-sectional study. In the full cross-sectional study experienced yogis will be matched on a number of variables with healthy controls not practicing any type of mind-body techniques. After screening, participants will be fitted with an ambulatory electrocardiography device (Holter monitor) for 24 hours to characterize their HRV in natural settings. They will also provide saliva samples at pre-determined intervals for seven consecutive days to measure cortisol, an index of the HPA axis function. Each subject will undergo two testing sessions. Session 1 will evaluate how participants anticipate and process warm and painful stimuli in certain and uncertain contexts by measuring perception while monitoring physiological responses such as respiration, heart rate, blood pressure, skin conductance and cortisol response. In session 2, functional magnetic resonance imaging (fMRI) will be used to assess potential differences in brain resting state activity between groups, as well as to document neural responses related to the anticipation and processing of warm and painfully hot stimuli in certain and uncertain contexts using a similar paradigm as in session 1. Once again, physiological monitoring will be performed. Anatomical MRI scans will be acquired for co-registration of the fMRI findings as well as to measure gray matter volume and cortical thickness differences between groups. Questionnaires evaluating the participants mental state and personality traits will be acquired throughout the sessions.

Outcome measures: Ratings of warm and painfully hot stimuli in certain and uncertain contexts will be compared between groups. Baseline HRV and cortisol levels will also be compared between groups. Functional and anatomical MRI data will be analyzed to examine differences between yogis and healthy volunteers for 1) gray matter volume and cortical thickness; 2) thermal anticipation and thermal-evoked activation patterns in certain and uncertain contexts; 3) functional connectivity during both anticipation and processing of thermal stimuli in certain and uncertain contexts; 4) resting state activity; and 5) functional connectivity during resting state. We will examine whether the behavioral, functional, or structural differences found are related to HPA axis function, autonomic function, personality traits and mental state.

ELIGIBILITY:
* FOR YOGA PRACTITIONERS:

You may qualify if you are:

* at least 30 years old
* an experienced yoga practitioner and practice regularly
* fluent in English
* right-handed
* in good health

You may not qualify if you:

* have a major medical condition
* suffer from chronic pain
* are pregnant or breast-feeding
* have a fear of enclosed spaces (claustrophobia)

FOR HEALTHY CONTROLS:

You may qualify if you are:

* at least 30 years old
* fluent in English
* right-handed
* in good health

You may not qualify if you:

* practice yoga, meditation, or martial arts
* have a major medical condition
* suffer from chronic pain
* are pregnant or breast-feeding

have a fear of enclosed spaces (claustrophobia)

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-01-27; Primary Completion 2015-10-19 (Actual); Study Completion 2016-10-12 (Actual)

PRIMARY OUTCOMES:
Pain perception (pain ratings) | 22 months

SECONDARY OUTCOMES:
Brain acivations, brain anatomy, autonomic response, cortisol | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Bushnell, Ph.D., Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fillingim RB. Individual differences in pain responses. Curr Rheumatol Rep. 2005 Oct;7(5):342-7. doi: 10.1007/s11926-005-0018-7. PMID 16174481
- [Background] Coghill RC, McHaffie JG, Yen YF. Neural correlates of interindividual differences in the subjective experience of pain. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8538-42. doi: 10.1073/pnas.1430684100. Epub 2003 Jun 24. PMID 12824463
- [Background] Villemure C, Bushnell CM. Cognitive modulation of pain: how do attention and emotion influence pain processing? Pain. 2002 Feb;95(3):195-199. doi: 10.1016/S0304-3959(02)00007-6. No abstract available. PMID 11839418